CLINICAL TRIAL: NCT00518648
Title: Reduction of Falls in the Elderly - Parkinson's Disease
Acronym: REFINE-PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: National Parkinson Foundation (Other)
Responsible Party: Dr. M. Munneke, UMC St Radboud, Neurology
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007_RP1.1
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Parkinson's Disease
Keywords: Accidental falls; Prevention; Treatment effectiveness
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Multifactorial fall prevention program
  Interventions: Other: Multifactorial fall prevention program
- II (Other): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Multifactorial fall prevention program — Individualised multifactorial fall prevention program containing PD-specific elements as well as generic elements
  Arms: I
Other: Usual care — Usual care
  Arms: II

SUMMARY:
The REFINE-PD study is a controlled trial embedded within a larger cluster controlled study (the IMPACT study). The study aims to investigate the efficacy of a multifactorial falls prevention program for patients with Parkinson's Disease (PD). This program contains PD-specific elements (e.g., optimizing dopaminergic therapy), plus a generic falls prevention program. The intervention will be tailored to each individual's specific risk profile for falls, as identified during detailed baseline examination.

DETAILED DESCRIPTION:
Falls and postural instability are common complications of advanced Parkinson's Disease (PD). Falls in PD often have devastating consequences, leading to a poor overall prognosis. In addition, falls in PD are associated with substantial medical expenses due to treatment of injuries and nursing home admission. The risk of falls in older PD patients is aggravated by "generic" age-related factors, such as sedative medication or poor vision. Observations on elderly persons without PD suggest that a multifactorial prevention program might be more effective. We propose to investigate the effectiveness of a multifactorial prevention program aimed at the prevention of falls in PD, which is based on disease-specific treatment strategies with demonstrated efficacy in PD, as well as prevention strategies with proven effectiveness for the general elderly population.

In this study an individualised multifactorial program aimed at the prevention of falls in PD containing PD-specific elements and a generic falls prevention program will be compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's Disease, diagnosed according to the Brain Bank criteria of the UK Parkinson's Society
* Regular control by the neurologist
* Living independently in the community
* Able to complete the trial questionnaires
* An increased risk for falling, defined as:

  * at least one fall in the preceding 12 months OR
  * recurrent (monthly) near falls in the preceding 12 months OR
  * fear of falling OR (iv) avoidance of activities due to fear of falling OR a combination of these findings

Exclusion Criteria:

* Atypical parkinsonian syndromes
* Hoehn and Yahr stage 5
* Severe cognitive impairment (MMSE < 24)
* Severe co-morbidity (e.g., cancer)
* Planned surgical procedure for PD within the intervention period
* Patients who have already visited the Multidisciplinary Assessment Center

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2007-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Incidence of falls | 8 months

SECONDARY OUTCOMES:
Number of fallers (secondary) | 8 months
Falls Efficacy Scale (tertiary) | 8 months
Unified Parkinson's Disease rating scale (UPDRS) Motor Examination (part III) (tertiary) | 4 months
Parkinson's Disease quality of life questionnaire (PDQL) (tertiary) | 8 months
Self-assessment Parkinson's Disease disability scale (SPDDS)(tertiary) | 8 months
Caregiver burden assessed with BELA-A-k, SF-36, and HADS (tertiary) | 8 months
Number of injurious falls (secondary) | 8 months
Number of patients with injurious falls (secondary) | 8 months
Freezing of gait (tertiary) | 8 months
Costs (secondary) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Marten Munneke, PhD, Principal Investigator — UMC St. Radboud; Bastiaan R. Bloem, MD, PhD, Principal Investigator — UMC St. Radboud; Marjolein A. van der Marck, MSc, Principal Investigator — UMC St. Radboud
Locations (6):
- Netherlands (6):
  - Ziekenhuis Groep Twente, Twenteborg Ziekenhuis, Almelo
  - Ziekenhuis Rijnstate, Arnhem
  - Wilhelmina Ziekenhuis Assen, Assen
  - Ziekenhuis Groep Twente, Streekziekenhuis Midden-Twente, Hengelo
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Canisius Wilhelmina Ziekenhuis, Nijmegen